CLINICAL TRIAL: NCT01025128
Title: Vitamin D Status in Males in Jerusalem Area and Its Correlation to Parathyroid Hormone (PTH) Level and Bone Mineral Density
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Metzger Muriel, MD, Clalit Health Services
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: K129/09
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Vitamin D Deficiency; Secondary Hyperparathyroidism; Osteomalacia
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism, Secondary; Osteomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- group A low D (Active Comparator): ultra-Orthodox clinics patients aged 18-39 with lowest vitamin D levels
  Interventions: Drug: 25 OH vitamin D
- group A high D (No Intervention): ultra-Orthodox clinics patients aged 18-39 with highest vitamin D levels
- group B low D (Active Comparator): mixed population clinics patients aged 18-39 with lowest vitamin D levels
  Interventions: Drug: 25 OH vitamin D
- group B high D (No Intervention): mixed population clinics patients aged 18-39 with highest vitamin D levels

INTERVENTIONS:
Drug: 25 OH vitamin D — oral supplementation of 25 OH vitamin D at dose of 2000 units/d for 3 months then 1000 units/d for 3 months
  Arms: group A low D; group B low D

SUMMARY:
Because of its high sun exposure, Israel was traditionally supposed to be protected from vitamin D deficiency, and the country food products hardly contain vitamin D supplements. However the Jerusalem ultra-Orthodox population, which constitutes a significant fraction of the city population, is at risk of developing vitamin D deficiency due to low sun exposure, as consequence of its dressing code covering most of the body and very limited time of outside activities. The investigators aim is to check whether vitamin D deficiency is found more frequently in the ultra-Orthodox male population in comparison to a non-ultra-Orthodox male population, and to study its eventual consequences. Correlation between vitamin D levels and PTH levels will be examined, according to age and to creatinine levels. Bone mineral density (BMD) will be evaluated in 2 selected subgroups of subjects (with lowest and highest vitamin D levels), and re-evaluated after 6 months of vitamin D supplementation in vitamin D-deficient subjects. An increase in BMD within 6 months would suggest osteomalacia as the main cause of low BMD in these subjects.

DETAILED DESCRIPTION:
Subjects:

The study will include 200 males aged 18-70, living in the Jerusalem area. Enrollment will be distributed among 8 clinics of the Clalit Health Services: 4 clinics located in predominantly ultra-Orthodox areas (group A) and 4 clinics located in mixed areas (Group B).

Each group of clinics will enroll 100 subjects as sub-defined:

Age 18-24: 30 patients (Groups A1 and B1) Age 25-39: 30 patients (Groups A2 and B2) Age 40-54: 20 patients (Groups A3 and B3) Age 55-70: 20 patients (Groups A4 and B4)

Study protocol:

Enrollment will be performed by the physicians participating in the study and the nurses working in the corresponding clinics, after advertisement of the study in the clinics.

Visit 1:

1. The subjects will receive information about the study aims and protocol and will sign an informed consent form.
2. Blood pressure, height and weight will be measured and BMI calculated.
3. The subjects will fill a questionnaire concerning their personal habits: dressing code, degree of sun exposure, physical activity, smoking, alcohol consumption, muscular pains and general fatigue.
4. The physician (co-investigator) signing the informed consent form will rule out subjects presenting pre-defined exclusion criteria.
5. Blood samples will be drawn for: calcium, phosphorus, PTH, 25 OH Vitamin D, 1,25 OH Vitamin D, magnesium, creatinine, alkaline phosphatase, albumin.
6. A urine sample will be collected for magnesium and calcium/creatinine ratio.

The subjects will receive the lab results by mail, with a recommendation to consult their family physician in order to receive treatment in case of vitamin D deficiency. (Vitamin D levels <20 ng/ml)

The subjects in the 18-39 age groups (Groups A1, A2, B1 and B2) will be classified according to their vitamin D levels. The 20 subjects presenting the highest vitamin D levels or with vitamin D level>30 ng/ml will constitute the "high D" group and the 40 subjects with the lowest vitamin D levels will constitute the "low D" group. (We expect the vitamin D levels to be above 30 ng/ml in the "high D" group and below 10 ng/ml in the "low D" groups, according to the results of our pilot study).

Subjects with vitamin D level>30 ng/ml or <10 ng/ml can be enrolled to the 60 patients of the "high D" and "low D " groups and will proceed to visits 2 and 3.

Visit 2:

60 subjects (20 from the "high D" group and 40 from the "low D" group) will undergo a bone mineral density examination in the Osteoporosis Center of Mount-Scopus Hadassah Hospital. All subjects with low vitamin D levels will receive a 6-month vitamin D supplementation of 2000 units per day for the first 12 weeks and of 1000 units per day for the next 12 weeks.

Visit 3:

The 60 subjects who underwent visit 2 will undergo visit 3 six months later.

1. The subjects will fill a questionnaire similar to the first one and detail their degree of compliance with vitamin D supplementation
2. Blood samples will be drawn for plasma levels of: calcium, phosphorus, magnesium, PTH, 25 OH vitamin D, 1,25 (OH)2 vitamin D, creatinine, alkaline phosphatase, albumin
3. A urine sample will be collected for magnesium and calcium/creatinine ratio.
4. A repeat bone mineral density examination will be performed in the Osteoporosis Center Mount-Scopus Hadassah Hospital

The subjects will receive their test results by mail with a recommendation to consult their family physician in case of persistent abnormal results.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-70
* If age below 40 must not be under any chronic medication

Exclusion Criteria:

* Medication: anti-convulsivants, non-topical steroids (past or present), anti-rejection medications
* Malabsorptive diseases (Crohn's disease, cystic fibrosis,Whipple' disease, s/p bariatric surgery)
* Morbid obesity (BMI above 35)
* Rheumatoid arthritis
* Liver failure
* Nephrotic syndrome
* Chronic kidney disease
* Genetic disorder
* Malignancy
* Primary hyperparathyroidism
* Granulomatous disease
* Hyperthyroidism
* Nephrolithiasis (present or past)
* S/P skin grafts surgery
* Mental disorder or cognitive disorder

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
plasma vitamin D level | 6 months

SECONDARY OUTCOMES:
bone mineral density before vitamin D supplementation | 8 months
plasma PTH level | 6 months
bone mineral density after vitamin D supplementation in vitamin D deficient subjects | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Metzger, MD, Principal Investigator — Clalit Health Services, Jerusalem, Israel; Anat Tsur, MD, Principal Investigator — Clalit Health Services, Jerusalem, Israel
Locations (1):
- Endocrinology Clinic, Clalit Health Services, Jerusalem, Israel